CLINICAL TRIAL: NCT05521139
Title: A Matched Case-control Study of Carbapenem Resistant and Carbapenem Sensitive Klebsiella Pneumoniae Infected Pyogenic Liver Abscess
Brief Title: Risk Factors for Pyogenic Liver Abscess With Carbapenem-resistant Klebsiella Pneumoniae: A Matched Case-control Study
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 202005055
Record Dates: First submitted 2022-08-29; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Liver Abscess
MeSH Terms: conditions — Liver Abscess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRKP-PLA: Klebsiella pneumoniae were isolated from pyogenic liver abscess patients' blood or pus and the antibiotic drug sensitivity results shows it is carbapenem-resistant Klebsiella pneumoniae.
  Interventions: Diagnostic Test: drug sensitivity results
- CSKP-PLA: Klebsiella pneumoniae were isolated from pyogenic liver abscess patients' blood or pus and the antibiotic drug sensitivity results shows it is carbapenem-sensitive Klebsiella pneumoniae.
  Interventions: Diagnostic Test: drug sensitivity results

INTERVENTIONS:
Diagnostic Test: drug sensitivity results — drug sensitivity results including the carbapenem-resistant Klebsiella pneumoniae and carbapenem-sensitive Klebsiella pneumoniae

SUMMARY:
Pyogenic liver abscess (PLA) is a complication of infectious disease, and the most common pathogen of PLA is Klebsiella pneumoniae, while PLA caused by Carbapenem-resistant Klebsiella pneumoniae (CRKP) has become a threat to public health. For achieving a better therapeutic outcome of CRKP related PLA, it is very important to figure out the basic characteristics and risk factors of CRKP-PLA.

A retrospective cohort study was performed in which 15 PLA patients carriage of K pneumoniae were screened at the Xiangya hospital of central south university (changsha, China). The colonization and clinical infection isolates were analyzed by antimicrobial susceptibility testing to identify CRKP. All admission patients diagnosed with PLA who developed CRKP were included, 5 adults PLA patients with CRKP infected and 10 adults PLA patients with Carbapenem sensitive Klebsiella pneumoniae (CSKP) infected were conducted. Univariate and multivariate logistic regression was carried out using a stepwise selection method to compare prognostic factors between CRKP and CSKP groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older. at least one positive culture reported by the clinical microbiology laboratory for CRKP or CSKP during the hospital length of stay.

Klebsiella pneumoniae were isolated and identified in the blood or pus with antibiotic drug sensitivity results.

Exclusion Criteria:

* Less than 18 years old. patients with missing data without a drug sensitivity results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age or older and at least one positive culture reported by the clinical microbiology laboratory for CRKP or CSKP during the hospital length of stay. Klebsiella pneumoniae were isolated and identified in the blood or pus with antibiotic drug sensitivity results.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
the survival rates | 2monthes

CONTACTS AND LOCATIONS:
Locations (1):
- Jinqing Liu, Changsha, China

IPD SHARING:
Plan to Share IPD: No